CLINICAL TRIAL: NCT00130559
Title: Does a Diagnostic Strategy Reduce Duration and Cost of Hospitalization in Patients With Acute Dyspnea? BASEL II Intensive Care Unit
Brief Title: B-type Natriuretic Peptide (BNP)-Guided Diagnostic Strategy in Intensive Care Unit (ICU) Patients With Respiratory Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: BASEL II - ICU; PP00B-102853/1; 04.061; 36/01
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Respiratory Insufficiency
Keywords: Respiratory failure; BNP
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: BNP guided diagnostics and initial therapy — BNP guided diagnostics and initial therapy

SUMMARY:
Heart failure is a common reason for respiratory failure in ICU patients. The rapid and accurate differentiation of heart failure from other causes of respiratory failure remains a clinical challenge. BNP levels are significantly higher in patients with congestive heart failure as compared to patients with respiratory failure due to other causes. Therefore, rapid measurement of BNP might be very helpful in establishing or excluding the diagnosis of heart failure in patients with respiratory failure in the ICU.

The aim is to test the hypothesis that a BNP guided diagnostic strategy would improve the evaluation and management of patients presenting with primary (on admission) or secondary (while in the ICU) respiratory failure in the ICU and thereby reduce total treatment time and total cost of treatment.

Primary endpoints are time to discharge and total cost of treatment. Secondary endpoints are ICU length of stay, ICU cost, in-hospital mortality, 30-day mortality, cost-effectiveness, 6 and 12 month mortality, 6 and 12 month dyspnea score.

DETAILED DESCRIPTION:
Background: Respiratory failure is not only the most important reason for admission of patients to a medical intensive care unit (ICU), but also a common reason for the deterioration of patients already treated in the ICU. It is a very serious condition associated with significant mortality. Heart failure is a common reason for respiratory failure in both circumstances. Unfortunately, the rapid and accurate differentiation of heart failure from other causes of respiratory failure in the ICU remains a clinical challenge. After evaluation of symptoms, physical examination, arterial blood gases, ECG, and chest x-ray, the clinician is often left with a considerable diagnostic uncertainty that results in misdiagnosis and delay in the initiation of appropriate therapy. In addition, misdiagnosis of heart failure causes morbidity, and increases total treatment time and treatment cost, because treatments for heart failure may be hazardous to patients with other conditions such as chronic obstructive pulmonary disease, and vice verse.

B-type natriuretic peptide (BNP) is a 32-amino acid polypeptide secreted from the cardiac ventricles in response to ventricular volume expansion and pressure overload. BNP levels are significantly higher in patients with congestive heart failure as compared to patients with respiratory failure due to other causes. Therefore, rapid measurement of BNP might be very helpful in establishing or excluding the diagnosis of heart failure in patients with respiratory failure in the ICU.

Aim: The aim is to test the hypothesis that a BNP guided diagnostic strategy would improve the evaluation and management of patients presenting with primary (on admission) or secondary (while in the ICU) respiratory failure in the ICU and thereby reduce total treatment time and total cost of treatment.

Endpoints: Primary endpoints: Time to discharge and total cost of treatment. Secondary endpoints: ICU length of stay, ICU cost, In-hospital mortality, 30-day mortality, cost-effectiveness, 6 and 12 month mortality, 6 and 12 month dyspnea score.

Patients and Methods: The trial is designed to enroll 286 patients presenting with primary (on admission) or secondary (while in the ICU) respiratory failure in the ICU. Patients will be randomly divided 1:1 into a clinical group using evaluation of patients according to local standards without the use of BNP (or other natriuretic peptides) and to a BNP group with early testing for BNP.

Expected results: The researchers hypothesize that a BNP guided diagnostic strategy will improve the evaluation and management of patients presenting with respiratory failure to the ICU and thereby reduce time to discharge and total cost of treatment.

Significance: If in fact, BNP testing could be shown to improve the evaluation and management of patients with respiratory failure in the ICU, this would represent a major advance in the clinical care of seriously ill patients, and as well, highlight the potential for considerable cost-saving. Accordingly, if this study would have a positive result and in fact demonstrate that a BNP guided diagnostic strategy reduces total treatment time and total cost of treatment, it would be the first randomized controlled trial demonstrating that a new diagnostic test improves the evaluation and management of ICU patients. Given the enormous expenses associated with intensive care, such a study seems overdue.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with primary or secondary respiratory failure in the ICU

Exclusion Criteria:

* Age <18 years
* Obvious traumatic cause
* Renal dysfunction (serum creatinine >250umol/l)
* Sepsis
* Cardiopulmonary reanimation within the last 12 hours
* Shock
* Respiratory insufficiency triggered during bronchoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2003-12; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Time to discharge | discharge
Total cost of treatment | until discharge

SECONDARY OUTCOMES:
ICU length of stay | discharge from ICU
ICU cost | until discharge from ICu
In-hospital mortality | discharge
30-day mortality | 30 days
cost-effectiveness | discharge
6 and 12 month mortality | 12 months
6 and 12 month dyspnea score | 12 months
Incidence/recognition of congestive heart failure (CHF) as a major cause of respiratory failure | discharge from ICU+
Incidence of diagnosed CHF as cause of respiratory failure in patients with COPD on ICU | discharge
Number of echo study performing during hospital stay | hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, Prof, Principal Investigator — University Hospital, Basel, Switzerland
Locations (6):
- Switzerland (6):
  - University Hospital Basel, Medical ICU, Basel, Canton of Basel-City
  - University Hospital Basel, Surgical ICU, Basel, Canton of Basel-City
  - Hospital of Interlaken, Interlaken, Canton of Bern
  - Hospital of Thun, Thun, Canton of Bern
  - Hospital of Luzern, Lucerne, Canton of Lucerne
  - Hospital of Solothurn, Solothurn, Canton of Solothurn

REFERENCES:
- [Background] Mueller C, Scholer A, Laule-Kilian K, Martina B, Schindler C, Buser P, Pfisterer M, Perruchoud AP. Use of B-type natriuretic peptide in the evaluation and management of acute dyspnea. N Engl J Med. 2004 Feb 12;350(7):647-54. doi: 10.1056/NEJMoa031681. PMID 14960741
- [Derived] Noveanu M, Breidthardt T, Reichlin T, Gayat E, Potocki M, Pargger H, Heise A, Meissner J, Twerenbold R, Muravitskaya N, Mebazaa A, Mueller C. Effect of oral beta-blocker on short and long-term mortality in patients with acute respiratory failure: results from the BASEL-II-ICU study. Crit Care. 2010;14(6):R198. doi: 10.1186/cc9317. Epub 2010 Nov 3. PMID 21047406
- [Derived] Noveanu M, Pargger H, Breidthardt T, Reichlin T, Schindler C, Heise A, Schoenenberger R, Manndorff P, Siegemund M, Mebazaa A, Marsch S, Mueller C. Use of B-type natriuretic peptide in the management of hypoxaemic respiratory failure. Eur J Heart Fail. 2011 Feb;13(2):154-62. doi: 10.1093/eurjhf/hfq188. Epub 2010 Oct 29. PMID 21036778
- See also: Related Info — http://www.dyspnea.ch